CLINICAL TRIAL: NCT02488317
Title: Empowering Patients On Choices for Renal Replacement Therapy (Aim 3)
Brief Title: Empowering Patients On Choices for Renal Replacement Therapy (Aim 3) (EPOCH-RRT)
Acronym: EPOCH-RRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: University of Michigan (Other); Henry Ford Health System (Other); National Kidney Foundation, United States (Other); American Association of Kidney Patients (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: 1109201303123
Record Dates: First submitted 2015-06-15; First posted 2015-07-02 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Hemodialysis; Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Other): These patients will receive the decision aid tool. Decision-making outcomes (e.g., self-efficacy) will be compared between patients who received and did not receive a decision aid. These arms were chosen because the current standard of care is for health care providers to discuss options with patients without using a decision aid.
  Interventions: Other: Decision Aid
- Control arm (No Intervention): These patients will not receive the decision aid tool and will be asked to test their knowledge without it. Decision-making outcomes (e.g., self-efficacy) will be compared between patients who received and did not receive a decision aid. These arms were chosen because the current standard of care is for health care providers to discuss options with patients without using a decision aid.

INTERVENTIONS:
Other: Decision Aid — Decision-making outcomes (e.g., self-efficacy) will be compared between patients who received and did not receive a decision aid. These arms were chosen because the current standard of care is for health care providers to discuss options with patients without using a decision aid.
  Arms: Intervention arm

SUMMARY:
Empowering Patients On Choices for Renal Replacement Therapy (EPOCH-RRT) study seeks to identify factors that matter the most to patients with kidney disease and study how they are impacted by different types of dialysis. The inclusion of patients, caregivers, and patient advocacy organizations as research partners will assure that the study addresses questions of greatest relevance to patients facing the need for dialysis.

For Aim 3, the investigators are going to compare measures related to the decision-making process between patients receiving and not receiving a decision aid focusing on Peritoneal Dialysis and Hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Speaks English
* Has access to the internet

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Tentori, MD, MS, Principal Investigator — Arbor Research Collaborative for Health
Locations (1):
- Arbor Research Collaborative for Health, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Subramanian L, Zhao J, Zee J, Knaus M, Fagerlin A, Perry E, Swartz J, McCall M, Bryant N, Tentori F. Use of a Decision Aid for Patients Considering Peritoneal Dialysis and In-Center Hemodialysis: A Randomized Controlled Trial. Am J Kidney Dis. 2019 Sep;74(3):351-360. doi: 10.1053/j.ajkd.2019.01.030. Epub 2019 Apr 4. PMID 30954312

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: These patients will not receive the decision aid tool and will be asked to test their knowledge without it. Decision-making outcomes (e.g., self-efficacy) will be compared between patients who received and did not receive a decision aid. These arms were chosen because the current standard of care is for health care providers to discuss options with patients without using a decision aid.
  Decision Aid: Decision-making outcomes (e.g., self-efficacy) will be compared between patients who received and did not receive a decision aid. These arms were chosen because the current standard of care is for health care providers to discuss options with patients without using a decision aid.
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 117 | 117
Completed | 63 | 70
Not Completed | 54 | 47

BASELINE CHARACTERISTICS:
Population: Baseline information was collected for 140, but only 133 participants completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 45 | 88
  >=65 years | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.16 (14.59) | 59.44 (14.16) | 59.30 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 30 | 35 | 65
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Preference for Shared Decision Making
Description: Measured using the scale from Degner, L. F., Sloan, J. A., & Venkatesh, P. (1996). The Control Preferences Scale. The Canadian journal of nursing research= Revue canadienne de recherche en sciences infirmieres, 29(3), 21-43. The CPS is a clinically relevant, easily administered, valid, and reliable measure of preferred roles in health-care decision-making. A pick-one approach was used to identify patient preference for an active, passive or collaborative role in dialysis treatment decision making.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Intervention Pre-test: Intervention arm responses prior to accessing the decision aid (N=70)
- Intervention Post-test: Intervention arm responses after accessing the decision aid (N=63)
- Control: Control arm with no decision aid.
Arm/Group | Intervention Pre-test | Intervention Post-test | Control
Number analyzed (Participants) | 70 | 63 | 70
participants
  My doctor(s) and I will decide together | 22 | 19 | 35
  I will decide after considering Dr's opinion | 44 | 38 | 35
  My doctor will decide with little input from me | 1 | 0 | 0
  My doctor will decide but will consider my opinion | 1 | 1 | 0
  I will decide with little input from Dr. | 2 | 5 | 0

2. Primary Outcome: Decisional Conflict
Description: Measured using the scale from O'Connor, Annette M. "Validation of a Decisional Conflict Scale." Medical Decision Making 15, no. 1 (February 1, 1995): 25-30. 16 item scale, responses to each statement are scored from 1 (strongly agree) to 5 (strongly disagree), with negative statements having reverse scoring; thus high scores indicate higher decisional conflict. Mean score per participant is calculated across all items, subtract by 1 and multiplied by 25. Score range= 0-100. Mean scores across all participants in each arm are reported.
Time Frame: 6 months
Population: All participants who completed the questionnaire were included in these analyses.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 63 | 70
scores on a scale
  Intervention pre-test | 43.6 (15.9) | 42.5 (17.1)
  Intervention post-test | 29.1 (13.7) | 42.5 (17.1)

3. Primary Outcome: Decision Self-efficacy
Description: Measured through the scale found in Decision Self-Efficacy Ottawa: Ottawa Hospital Research Institute; © 1995 Available from: http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf O'Connor 1995 Items are scored 0(not at all confident) to 4 (very confident). Scores are summed across 10 items, divided by 10 and multiplied by 25. Scores range from 0-100. A score of 0 means "extremely low self efficacy" and a score of 100 means "extremely high self efficacy".
Time Frame: 6 months
Population: All participants who completed the questionnaire were included in these analyses.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 63 | 70
scores on a scale
  Intervention pre-test | 82.8 (18.0) | 79.9 (17.6)
  Intervention post-test | 82.0 (18.4) | 79.9 (17.6)

4. Primary Outcome: Knowledge
Description: Measured using scale from Cavanaugh K"Patient Dialysis Knowledge Is Associated with Permanent Arteriovenous Access Use in Chronic Hemodialysis." Clinical Journal of the American Society of Nephrology 4, no. 5: 950-56) Multiple choice questions with one correct answer per questions. Number of correct questions reported as a percentage of total number of questions (23).
Time Frame: 6 months
Population: All participants who completed the questionnaire were included in these analyses.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 63 | 70
scores on a scale | 90.3 (11.9) | 76.5 (15.3)

5. Primary Outcome: Preparation for Decision Making
Description: Measured using Bennett, Carol, "Validation of a Preparation for Decision Making Scale." Patient Education and Counseling 78, no. 1: 130-33 10 item scale, each item scored from 1 (not at all) to 5 (a great deal). items are summed and scored, converted to a 0-100 scale by subtracting 1 from the summed score and multiplying by 25. Higher scores indicate higher perceived level of preparation for decision making.
Time Frame: 6 months
Population: This was a comparison of the intervention group before and after using the decision aid to assess its impact on preparing the participant for decision making. The question was therefore not administered to the control group since a similar pre/post comparison could not be tested in this group that was not exposed to the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Post-test: Intervention arm after reviewing the decision aid
Arm/Group | Intervention Post-test
Number analyzed (Participants) | 63
units on a scale | 76.39 (18.86)

ADVERSE EVENTS:
Arm/Group | Intervention Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/117
Other Adverse Events (participants affected / at risk) | 0/117 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No